CLINICAL TRIAL: NCT06634719
Title: A Prospective Multicenter Safety and Feasibility Study of the Juveena Hydrogel System for Use for Temporary Control of Chronic Ovulatory Heavy Menstrual Bleeding (HMB)
Brief Title: Juveena Hydrogel System Feasibility Study for Heavy Menstrual Bleeding (HMB)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rejoni Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: REJ-CT-0008
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Intervention Model Description: Women with HMB
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Juveena Hydrogel System (Experimental): One time instillation of the Juveena Hydrogel into the uterine cavity.
  Interventions: Device: Juveena Hydrogel System

INTERVENTIONS:
Device: Juveena Hydrogel System — The Juveena Hydrogel System is a single-use device that is instilled into the endometrial cavity as a liquid and sets up as a gel intrauterine tamponade within seconds.

SUMMARY:
This is a prospective, multicenter, single-arm interventional feasibility study to evaluate the safety and feasibility of the Juveena Hydrogel System for temporary control of heavy menstrual bleeding (HMB) in women with a history of chronic ovulatory HMB.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm interventional feasibility study to evaluate the safety and feasibility of the Juveena Hydrogel System (HS) for temporary control of heavy menstrual bleeding (HMB) in women with a history of chronic ovulatory HMB.

Consenting subjects will be screened for eligibility and will have a baseline evaluation, including medical and gynecological history, and characterization of their menstrual cycle.

Eligible subjects will be tentatively scheduled for Juveena HS treatment, aiming for device placement no later than 3 days into the anticipated HMB component of their menstrual cycle. Subjects will be provided access to and instructions for populating a diary based on the Mansfield-Voda-Jorgensen (MVJ) menstrual bleeding scale, to be started on day 1 of the index menstrual period. On treatment day, eligibility will be confirmed (including confirmation of HMB and a negative urine pregnancy test) and an MVJ score documented pre- and post-treatment. Phone visits will be conducted post-treatment Days 1, 14 and 56. Clinic visits will be conducted post-treatment on Day 7 and Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 to 45 years inclusive seeking treatment for HMB
2. Recent history (within the last 3 months) of repeat periods of HMB that adversely affects quality of life (Modified SAMANTA score ≥4 and comprises at least three consecutive days of HMB, see Appendix 2).(23).
3. Historical menstrual pattern with at least 3 days (72 hours) of HMB as determined by retrospective MVJ Bleeding scale score of ≥5for prior cycle.
4. Menses frequency (24-38 days) based on subjectparticipant reporting.
5. Menses regularity - shortest to longest period is ≤8 days based on subjectparticipant reporting.
6. Actively experiencing heavy to very heavy menstrual bleeding (HMB) at the time of the Juveena HS treatment, i.e., MVJ score of ≥5 (treatment must be performed no later than Day 3 of the index period).
7. HMB refractory to hormone therapy, hormone therapy contraindicated, or subjectparticipant does not wish to continue hormone therapy.
8. The subjectparticipant is literate and clearly demonstrates an understanding of how to complete the MVJ Scale and other patient-reported outcomes.
9. Able and willing to comply with the study protocol and agrees to the following during participation in the study:

   1. Use an effective non-hormonal method of birth control until the Day 28 visit. Acceptable methods of birth control for use in this study are abstinence and barrier contraceptives (e.g. condom)
   2. No initiation or continuation of hormone use (including contraception) or any other medical intervention for bleeding until after the Day 28 visit (unless clinically necessary, e.g., the subjectparticipant becomes hemodynamically unstable)
   3. Attends the follow-up examexams and completion of electronic diaries via a secured internet website (subject must have internet accesscompletes the MVJ scale and will be trained on how to use the eDiary)other patient-reported outcomes per the schedule of events
10. Demonstrates understanding of the study and signs the written informed consent form.

Exclusion Criteria:

1. Pregnancy and/or breastfeeding within the past 3 months or planning to become pregnant during the duration of this study.
2. Currently using an intrauterine device (IUD) or has undergone removal within the last 2 menstrual cycles.
3. Dysmenorrhea of a severity that, in the opinion of the investigator, precludes participation in the study.
4. Hemoglobin of < 8 g/dL at the time of screening.
5. Suspected or known malignancy or premalignant condition of the uterus including the cervix
6. Active pelvic infection.
7. Active sexually transmitted disease (STD) at the time of treatment (STD testing to be performed)
8. Presence of bacteremia, sepsis, or other active systemic infection
9. Currently on anticoagulants
10. History of allergies to PEG or FD&C Blue#1 dye
11. Planning to undergo surgery or other treatments for HMB during the study period (i.e., 8 weeks post-hydrogel instillation).
12. AUB-L sm with a Type 0 or 1 leiomyoma > 1 cm
13. AUB-P (Polyp) > 2 cm in maximum dimension based on ultrasound, hysteroscopy, or MRI performed within prior 6 months.
14. AUB-O, Irregular menstrual cycles (cycle length variability >7 days length)
15. AUB-C (coagulopathy or bleeding disorder)
16. Any patient who is currently participating or considering participation in any other research of an investigational drug or device. Does not include observational studies
17. Any general health, mental health, or social situation which, in the opinion of the investigator, could represent an increased risk for the patient or the ability of the patient to complete study requirements.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with history of chronic HMB
Enrollment: 7 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | Within 7 days post-treatment
  Feasibility for invoking a tamponade effect

OTHER OUTCOMES:
Bleeding Control | Within 7 days post-treatment
  The proportion of subjects achieving bleeding control defined as none or spotting (MVJ ≤1)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Arizona Gynecology Consultants, Phoenix, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Rubino OB/GYN (Axia Women's Health), West Orange, New Jersey
  - Seven Hills Clinical Research Group, LLC, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No